CLINICAL TRIAL: NCT02369328
Title: Multimodal MRI Study of Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A01532-45
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: STROKE
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- multimodal MRI (Experimental): Multimodal MRI (including perfusion MRI, sodium MRI, resting-state functional MRI, high resolution anatomical MRI) and clinical evaluation will be carried on at the inclusion, after 24 hours, at 3 months and at 12 months for patients whom suffering stroke
  Interventions: Device: MULTIMODAL MRI
- multimocal MRI (Active Comparator): Multimodal MRI (including perfusion MRI, sodium MRI, resting-state functional MRI, high resolution anatomical MRI) and clinical evaluation will be carried on at the inclusion, after 24 hours, at 3 months and at 12 months for healthy subjects
  Interventions: Device: MULTIMODAL MRI

INTERVENTIONS:
Device: MULTIMODAL MRI — Multimodal MRI (including perfusion MRI, sodium MRI, resting-state functional MRI, high resolution anatomical MRI) will be carried on at the inclusion, after 24 hours, at 3 months and at 12 months and neurological clinical exam , rankin score, NIHSS

SUMMARY:
Stroke is the second most frequent causes of mortality in the word after cardiovascular disease and the most frequent cause of disability. The majority of strokes are ischemic (87%). Ischemic stroke may benefit from efficient therapy if the delay from stroke onset not exceeds 4H30 (intra-venous thrombolysis). In case of irreversible cerebral lesion, the long term functional recovery is largely dependent from the ability of the brain to reorganize. Conventional magnetic resonance imaging represents the most sensitive tool to diagnose stroke at the acute phase. However, up to now, no imaging tool is available to determine the time of stroke onset. Moreover, no imaging tool is available to precisely quantify the functional and structural plasticity mechanisms occurring after stroke. The main objective of the present study is to test the accuracy of sodium MRI to determine the time of stroke onset. The secondary objectives of the study are to determine the ability of non-conventional MRI techniques to quantify the degree of tissue damage and brain reorganization after stroke. Thirty patients will be included during the first 24 hours after stroke onset. Multimodal MRI (including perfusion MRI, sodium MRI, resting-state functional MRI, high resolution anatomical MRI) and clinical evaluation will be carried on at the inclusion, after 24 hours, at 3 months and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

- Patient having presented a cerebral infarct beforehand confirmed by the brain imaging

* Patient having presented a cerebral infarct the hour of the beginning of which is known with certainty and dating less than 24 hours
* Patient having presented a cerebral infarct the area(extent) of which is superior to 1,5 ml

Exclusion Criteria:

* Patients presenting the usual contraindications to the MRI (pacemaker, agitation, metallic brightness, claustrophobia etc.)
* Patients presenting a risk of not compliance to the examination: disorders(confusions) of the elementary understanding, the confusion, the involuntary movements, the bad tolerance of the prolonged dorsal decubitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The time of stroke onset | 3 years
  The main objective of the present study is to test the accuracy of sodium MRI to determine the time of stroke onset

SECONDARY OUTCOMES:
The degree of tissue damage and brain reorganization after stroke | 3 years
  The secondary objectives of the study are to determine the ability of non-conventional MRI techniques to quantify the degree of tissue damage and brain reorganization after stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, Marseille, France